CLINICAL TRIAL: NCT00560235
Title: A Phase 1/Phase 2 Study Of CP-751,871 In Patients With Relapsed And/Or Refractory Ewing's Sarcoma Family Of Tumors
Brief Title: Study Of CP-751,871 In Patients With Ewing's Sarcoma Family Of Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021020
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Ewing's Sarcoma Family of Tumors
MeSH Terms: interventions — figitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CP-751,871

INTERVENTIONS:
Drug: CP-751,871 — Final dose 30 mg/kg IV on Day 1 of each 28 day cycle until either progression or toxicity

SUMMARY:
Define the efficacy of CP-751,871 in patients with Ewing's sarcoma family of tumors

ELIGIBILITY:
Inclusion Criteria:

* Ewing's family of tumors
* Current disease state for which there is no curative therapy

Exclusion Criteria:

* Prior anti-IGF-1R therapy
* Concurrent treatment with other anti-cancer agents

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (9):
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Australia (2):
  - Pfizer Investigational Site, Brisbane, Queensland
  - Pfizer Investigational Site, Parkville, Victoria
- Pfizer Investigational Site, São Paulo, São Paulo, Brazil
- Pfizer Investigational Site, Toronto, Ontario, Canada
- Pfizer Investigational Site, Providencia, Santiago, RM, Chile
- France (4):
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Villejuif
- Germany (4):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
- Israel (2):
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Petah Tikva
- Italy (3):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Torino
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Esplugues de Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
- United Kingdom (3):
  - Pfizer Investigational Site, Sutton, Surrey
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Oxford

REFERENCES:
- [Derived] Juergens H, Daw NC, Geoerger B, Ferrari S, Villarroel M, Aerts I, Whelan J, Dirksen U, Hixon ML, Yin D, Wang T, Green S, Paccagnella L, Gualberto A. Preliminary efficacy of the anti-insulin-like growth factor type 1 receptor antibody figitumumab in patients with refractory Ewing sarcoma. J Clin Oncol. 2011 Dec 1;29(34):4534-40. doi: 10.1200/JCO.2010.33.0670. Epub 2011 Oct 24. PMID 22025154
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited separately for Phase 1 and Phase 2. A total of 138 participants were assigned to received study treatment (31 participants for Phase 1 and 107 participants for Phase 2).
Groups:
- Figitumumab Dose Escalation (Phase 1): Figitumumab 20 milligrams per kilogram (mg/kg) intravenous (IV) administered every 4 weeks (1 cycle). If no dose-limiting toxicity (DLT) was identified in the 20-mg/kg cohort, dose escalation proceeded to 30-mg/kg. Oral rapamycin at 2 to 4 mg/day could have been added as salvage therapy.
- Figitumumab Dose Extension (Phase 1B): Figitumumab 20 mg/kg or 30 mg/kg IV administered every 4 weeks (1 cycle). Oral rapamycin at 2 to 4 mg/day could have been added as salvage therapy.
- Figitumumab 30 mg/kg (Phase 2): Figitumumab 30 mg/kg IV administered every 4 weeks (1 cycle) for up to 12 cycles, unless unacceptable toxicity or participant withdrawal. Oral rapamycin at 2 to 4 mg/day could have been added as salvage therapy.
Period: Phase 1
Arm/Group | Figitumumab Dose Escalation (Phase 1) | Figitumumab Dose Extension (Phase 1B) | Figitumumab 30 mg/kg (Phase 2)
Started | 10 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 8 | 0 | 0
Not completed — Discontinued | 8 | 0 | 0
Period: Phase 1B
Arm/Group | Figitumumab Dose Escalation (Phase 1) | Figitumumab Dose Extension (Phase 1B) | Figitumumab 30 mg/kg (Phase 2)
Started | 0 | 21 | 0
Completed | 0 | 2 | 0
Not Completed | 0 | 19 | 0
Not completed — Discontinued | 0 | 19 | 0
Period: Phase 2
Arm/Group | Figitumumab Dose Escalation (Phase 1) | Figitumumab Dose Extension (Phase 1B) | Figitumumab 30 mg/kg (Phase 2)
Started | 0 | 0 | 107
Completed | 0 | 0 | 10
Not Completed | 0 | 0 | 97
Not completed — Discontinued | 0 | 0 | 96
Not completed — Ongoing at Date of Cut-Off | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Figitumumab Dose Escalation (Phase 1) | Figitumumab Dose Extension (Phase 1B) | Figitumumab 30 mg/kg (Phase 2) | Total
Number analyzed (Participants) | 10 | 21 | 107 | 138
Age, Customized [Number; unit: participants]
  10 to <13 years | 2 | 3 | 17 | 22
  13 to <=18 years | 8 | 18 | 30 | 56
  18 to <30 years | 0 | 0 | 43 | 43
  30 to <41 years | 0 | 0 | 10 | 10
  >=41 years | 0 | 0 | 7 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 40 | 51
  Male | 6 | 14 | 67 | 87

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as complete disappearance of all target and non-target disease and no new lesions. PR was defined as ≥30% decrease under baseline of the sum of diameters of all target lesions.
Time Frame: Baseline and every cycle (4 weeks), for up to 6 cycles
Population: All enrolled participants with Ewing's sarcoma family of tumors (ESFT) and who started treatment with figitumumab; number of evaluable participants at data cut-off.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Figitumumab 30 mg/kg (Phase 2)
Number analyzed (Participants) | 106
percentage of participants | 14.2 [8.1 to 22.3]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was the time in months from start date to date of first documentation of progression, death due to any cause or symptomatic deterioration (global deterioration of health status requiring discontinuation of treatment).
Time Frame: Baseline and every cycle (4 weeks), until progression or death
Population: All enrolled participants with ESFT and who started treatment with figitumumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab 30 mg/kg (Phase 2)
Number analyzed (Participants) | 107
months | 1.9 [1.8 to 2.1]

3. Secondary Outcome: Overall Survival (OS)
Description: Time in months from enrollment to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: Baseline and every 2 cycles (8 weeks), until death or up to 6 cycles after date of enrollment
Population: All enrolled participants with ESFT and who started treatment with figitumumab.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Figitumumab 30 mg/kg (Phase 2)
Number analyzed (Participants) | 107
months | 8.9 [7.2 to 10.8]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Cycle 1 and Cycle 5: 1 hour post-infusion on Day 1
Population: The pharmacokinetic (PK) analysis set included all enrolled participants who started treatment and who had sufficient samples to provide interpretable results; n=number of participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per liter (mg/L)
Groups:
- Figitumumab 20 mg/kg Dose Escalation (Phase 1): Figitumumab 20 mg/kg IV was administered every 4 weeks (1 cycle).
- Figitumumab 30 mg/kg Dose Escalation (Phase 1); Figitumumab 30 mg/kg Dose Extension (Phase 1B): Figitumumab 30 mg/kg IV was administered every 4 weeks (1 cycle).
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B)
Number analyzed (Participants) | 4 | 6 | 21
milligrams per liter (mg/L)
  Cycle 1 (n=4, 6, 21) | 513.2 (42) [lower limit 42] | 1075 (21) [lower limit 21] | 975.6 (26) [lower limit 26]
  Cycle 5 (n=2, 2, 8) | 729.0 (47) [lower limit 47] | 1133 (9) [lower limit 9] | 1043 (47) [lower limit 47]

5. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Description: Cmin is the concentration at the end of treatment cycle (next cycle predose).
Time Frame: Cycle 6: predose on Day 1
Population: The PK analysis set included all enrolled participants who started treatment and who had sufficient samples to provide interpretable results; number of participants evaluated for measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B)
Number analyzed (Participants) | 1 | 1 | 7
mg/L | 389.0 | 345.0 | 283.6 (53) [lower limit 53]

6. Secondary Outcome: Plasma Concentration at End of Infusion (Cendinf)
Time Frame: Cycle 1 Day 2 and Cycle 5 Day 1
Population: The PK analysis set included all enrolled participants who started treatment and who had sufficient samples to provide interpretable results; n=number of participants evaluable for this measure at specified time points for each arm group, respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B)
Number analyzed (Participants) | 4 | 6 | 21
mg/L
  Cycle 1 (n=4, 6, 21) | 513.2 (42) [lower limit 42] | 1075 (21) [lower limit 21] | 975.6 (26) [lower limit 26]
  Cycle 5 (n=2, 2, 8) | 729.0 (47) [lower limit 47] | 1133 (9) [lower limit 9] | 1043 (47) [lower limit 47]

7. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: The dosing interval was 1 cycle (4 weeks) in this study.
Time Frame: Cycle 5: 1 hour post-infusion on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram*hour per liter (mg*hr/L)
Groups:
- Figitumumab 20 mg/kg Dose Escalation (Phase 1): Figitumumab 20 mg/kg IV administered every 4 weeks (1 cycle).
- Figitumumab 30 mg Dose Escalation (Phase 1): Figitumumab 30 mg/kg IV administered every 4 weeks (1 cycle).
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B)
Number analyzed (Participants) | 1 | 1 | 6
milligram*hour per liter (mg*hr/L) | 423000 | 475000 | 302900 (46) [lower limit 46]

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: AUClast is the area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: Cycle 1 and Cycle 5: 1 hour post-infusion on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*hr/L
Groups:
- Figitumumab 30 mg/kg Dose Escalation (Phase 1); Figitumumab 30 mg/kg Dose Extension (Phase 1B): Figitumumab 30 mg/kg IV administered every 4 weeks (1 cycle).
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B)
Number analyzed (Participants) | 4 | 6 | 21
mg*hr/L
  Cycle 1 (n=3, 5, 16) | 187200 (37) [lower limit 37] | 338800 (16) [lower limit 16] | 343000 (25) [lower limit 25]
  Cycle 5 (n=1, 1, 6) | 423000 (NA) [lower limit NA] — Geometric CV(%) not calculated as only 1 participant was evaluated. | 509000 (NA) [lower limit NA] — Geometric CV(%) not calculated as only 1 participant was evaluated. | 310800 (46) [lower limit 46]

9. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) Titer
Description: Number of participants with positive sample(s) in the ADA assay and in the neutralizing anti-drug antibodies (NAb) assay. An endpoint titer <6.64 corresponded to negative ADA category value.
Time Frame: Cycle 4 (predose on Day 1), 28 days after last dose (End-of-Treatment), and follow-up (approximately 150 days after last dose)
Population: All enrolled participants with ESFT and who started treatment with figitumumab. None of the serum samples were positive for ADAs following repeated administration of figitumumab, as indicated by an endpoint titer of <6.64.
Measure: Number; unit: participants
Arm/Group | Figitumumab 30 mg/kg (Phase 2)
Number analyzed (Participants) | 107
participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Figitumumab 20 mg/kg + Rapamycin Dose Escalation (Phase 1): Figitumumab 20 mg/kg IV was administered every 4 weeks (1 cycle). As optional salvage therapy for disease progression, oral rapamycin at 2 to 4 mg/day was administered in combination with figitumumab.
- Figitumumab 30 mg/kg + Rapamycin Dose Escalation (Phase 1); Figitumumab 30 mg/kg + Rapamycin Dose Extension (Phase 1B); Figitumumab 30 mg/kg + Rapamycin (Phase 2): Figitumumab 30 mg/kg IV was administered every 4 weeks (1 cycle). As optional salvage therapy for disease progression, oral rapamycin at 2 to 4 mg/day was administered in combination with figitumumab.
- Figitumumab 30mg/kg (Phase 2): Figitumumab 30 mg/kg IV was administered every 4 weeks (1 cycle) until unacceptable toxicity or participant withdrawal, for up to 6 cycles.
Arm/Group | Figitumumab 20 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) | Figitumumab 30 mg/kg Dose Extension (Phase 1B) | Figitumumab 20 mg/kg + Rapamycin Dose Escalation (Phase 1) | Figitumumab 30 mg/kg + Rapamycin Dose Escalation (Phase 1) | Figitumumab 30 mg/kg + Rapamycin Dose Extension (Phase 1B) | Figitumumab 30mg/kg (Phase 2) | Figitumumab 30 mg/kg + Rapamycin (Phase 2)
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/6 | 10/21 | 0/1 | 3/4 | 7/9 | 47/107 | 16/29
Other Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 19/21 | 1/1 | 3/4 | 9/9 | 99/107 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg Dose Escalation (Phase 1) (N=4) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) (N=6) | Figitumumab 30 mg/kg Dose Extension (Phase 1B) (N=21) | Figitumumab 20 mg/kg + Rapamycin Dose Escalation (Phase 1) (N=1) | Figitumumab 30 mg/kg + Rapamycin Dose Escalation (Phase 1) (N=4) | Figitumumab 30 mg/kg + Rapamycin Dose Extension (Phase 1B) (N=9) | Figitumumab 30mg/kg (Phase 2) (N=107) | Figitumumab 30 mg/kg + Rapamycin (Phase 2) (N=29)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 1 | 6 | 0 | 2 | 3 | 22 | 12
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Acinetobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 20 mg/kg Dose Escalation (Phase 1) (N=4) | Figitumumab 30 mg/kg Dose Escalation (Phase 1) (N=6) | Figitumumab 30 mg/kg Dose Extension (Phase 1B) (N=21) | Figitumumab 20 mg/kg + Rapamycin Dose Escalation (Phase 1) (N=1) | Figitumumab 30 mg/kg + Rapamycin Dose Escalation (Phase 1) (N=4) | Figitumumab 30 mg/kg + Rapamycin Dose Extension (Phase 1B) (N=9) | Figitumumab 30mg/kg (Phase 2) (N=107) | Figitumumab 30 mg/kg + Rapamycin (Phase 2) (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 14 | 9
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 13 | 2
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Eye movement disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 5 | 0 | 0 | 0 | 15 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 8 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 5 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 20 | 9
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 5 | 0 | 0 | 2 | 15 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 6 | 0 | 0 | 2 | 16 | 9
Retching (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0 | 2 | 3 | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 8 | 0 | 0 | 3 | 17 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 13 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 5 | 0 | 0 | 5 | 15 | 4
Fatigue (General disorders) | 1 | 2 | 4 | 0 | 0 | 2 | 27 | 10
General physical health deterioration (General disorders) | 0 | 0 | 2 | 0 | 1 | 5 | 4 | 5
Impaired healing (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 3
Pain (General disorders) | 0 | 2 | 1 | 0 | 1 | 3 | 5 | 4
Pyrexia (General disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 13 | 7
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 3
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 6 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breath sounds (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2 | 0 | 0 | 2 | 11 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 4 | 0 | 0 | 4 | 13 | 10
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 2 | 22 | 13
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 12 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 0 | 4 | 11 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 17 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 4 | 3
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 10 | 0 | 0 | 0 | 20 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 3 | 11 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 2 | 9 | 3
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1
Headache (Nervous system disorders) | 0 | 1 | 4 | 0 | 0 | 2 | 19 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 2 | 17 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 4 | 16 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 3 | 8 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 5 | 3
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 7 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 6 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amputation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scleral hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth discolouration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucous membrane disorder (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papilloma viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Right ventricular systolic pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Fear (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Perineal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immobile (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Vasodilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.